CLINICAL TRIAL: NCT02625337
Title: Phase 2 Study Comparing Pembrolizumab With Intermittent/Short-term Dual MAPK Pathway Inhibition Plus Pembrolizumab in Patients Harboring the BRAFV600 Mutation
Brief Title: Study Comparing Pembrolizumab With Dual MAPK Pathway Inhibition Plus Pembrolizumab in Melanoma Patients
Acronym: IMPemBra
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N15IMP
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; dabrafenib; trametinib; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pembrolizumab mono (Active Comparator): Pembrolizumab monotherapy
  Interventions: Drug: Pembrolizumab; Procedure: Biopsy; Procedure: Blood taking
- Pembrolizumab with dabrafenib+trametinib short (Experimental): Pembrolizumab combined with a short scheme of dabrafenib+trametinib
  Interventions: Drug: Pembrolizumab; Drug: Dabrafenib; Drug: Trametinib; Procedure: Biopsy; Procedure: Blood taking
- Pembrolizumab with dabrafenib+trametinib intermediate (Experimental): Pembrolizumab combined with an intermediate scheme of dabrafenib+trametinib
  Interventions: Drug: Pembrolizumab; Drug: Dabrafenib; Drug: Trametinib; Procedure: Biopsy; Procedure: Blood taking
- Pembrolizumab with dabrafenib+trametinib long (Experimental): Pembrolizumab combined with a long scheme of dabrafenib+trametinib
  Interventions: Drug: Pembrolizumab; Drug: Dabrafenib; Drug: Trametinib; Procedure: Biopsy; Procedure: Blood taking

INTERVENTIONS:
Drug: Pembrolizumab
Drug: Dabrafenib
  Arms: Pembrolizumab with dabrafenib+trametinib intermediate; Pembrolizumab with dabrafenib+trametinib long; Pembrolizumab with dabrafenib+trametinib short
Drug: Trametinib
  Arms: Pembrolizumab with dabrafenib+trametinib intermediate; Pembrolizumab with dabrafenib+trametinib long; Pembrolizumab with dabrafenib+trametinib short
Procedure: Biopsy — Biopsies will be taken during screening, before randomization, at week 8 (only arm 2-4) after 12 weeks, at week 18 and if PD.
Procedure: Blood taking — Blood will be taken for PBMCs during screening (twice), before randomization, at weeks 12 at week 18 and if PD.

SUMMARY:
This is a Phase 2 trial consisting of 24 patients receiving the combination of dabrafenib + trametinib + pembrolizumab in 3 different dosing schemes and 8 patients receiving pembrolizumab standard monotherapy. All patients start with pembrolizumab standard therapy for 6 weeks and will then be randomized to continue pembrolizumab monotherapy or to receive additional intermitted/short-term dabrafenib + trametinib.

Stratification will be baseline LDH level and baseline PD-L1 expression.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* World Health Organization (WHO) Performance Status 0-2
* Histologically/cytologically confirmed stage IV BRAF V600E or K metastatic melanoma
* Measurable disease according to RECIST 1.1
* At least one easy accessible lesion (s.c., lymph node) that can be repeatedly biopsied
* Patient willing to undergo triple tumor biopsies during screening, at week 6, week 8 (cohorts 2-4 only), week 12, at week 18, and in case of disease progression.
* No prior immunotherapy targeting PD-1 or PD-L1 (CTLA-4 targeting therapy is allowed)
* No prior BRAF and/or MEK targeting therapy
* No immunosuppressive medications
* Screening laboratory values must meet the following criteria:

WBC ≥ 2.0x109/L, Neutrophils ≥ 1.0x109/L, Platelets ≥ 100 x109/L, Hemoglobin ≥ 5.0 mmol/L Creatinine ≤ 2x ULN AST, ALT ≤ 2.5 x ULN (≤5 x ULN for patients with liver metastases) Bilirubin ≤2 X ULN

* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Women of child bearing potential must agree to use a reliable form of contraceptive during the study treatment period and for at least 120 days following the last dose of study drug
* Men must agree to the use of male contraception during the study Treatment Period and for at least 180 days after the last dose of study drug.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from this study:

* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Presence of symptomatic brain or leptomeningeal metastases; patients with asymptomatic brain metastases detected during screening for this study are allowed to participate in this study
* Prior PD-1/PD-L1 targeting immunotherapy
* Has an active automimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Known history of Human Immunodeficiency Virus;
* Active infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA);
* Has active tuberculosis
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy. Patients that have had another malignancy, but are free of tumor for more than 2 years are allowed for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety of different schemes of continuous/intermittent dabrafenib+trametinib during treatment with pembrolizumab as compared to pembrolizumab monotherapy as measured by SUSARs. | 18 weeks from baseline
  Safety as measured by SUSARs during treatment week 0 till week 18.
Feasibility of different schemes of continuous/intermittent dabrafenib+trametinib during treatment with pembrolizumab as compared to pembrolizumab monotherapy as measured by adherence to the timelines in the study protocol. | 18 weeks from baseline.
  Feasibility as measured by adherence to the timelines in the study protocol (week 0 till week 18).
The immune-activating capacity of different schemes of continuous/intermittent dabrafenib+trametinib during treatment with pembrolizumab as compared to pembrolizumab monotherapy | 18 weeks from baseline.
  Readout will be the alterations in magnitude or breadth of the self-antigen specific T cell responses in the time interval pre-treatment to week 18 intrapatient, and interpatient, pembrolizumab only (cohort 1) versus pembrolizumab plus intermittent dabrafenib/ trametinib (cohorts 2-4). To this purpose, we will analyze melanoma antigen-specific T cells responses by HLA-A2-restricted MHC-tetramer staining.

SECONDARY OUTCOMES:
To determine rates of response at week 6, 12, week 18. | Screening, week 6, 12 and 18
  Rates of response at week 6, week 12, week 18 according to RECIST 1.1 criteria
To determine progression-free survival starting from randomization. | From randomisation until PD, median 10 months.
  Progression-free survival (PFS) starting from randomization to progression using RECIST 1.1 criteria.
Long-term toxicities of intermittent dabrafenib + trametinib during treatment with pembrolizumab as compared to pembrolizumab monotherapy | From beyond week 18, up to 2 years follow-up.
  Rate and type of late adverse events

OTHER OUTCOMES:
To describe time to progression beginning from week 12 (cohorts 2-4). | Randomisation until week 12.
  As the short addition of dabrafenib+trametinib will induce for short time tumor regressions we will analyze cohorts 2-4 with a second baseline, namely the end of the targeted therapy at week 12, for progression free survival using to RECIST 1.1
Changes of immune parameters within the tumor. | 18 weeks from baseline.
  In addition to the primary readout (broadening of the melanoma-specific T cell response in peripheral blood), we will analyze the effect of the different therapy schemes on tumor immune cell infiltration (IHC for CD3, CD4, CD8, CD68, FoxP3, PD-L1, PD-L2, PD-1, CD11b, HLA).

CONTACTS AND LOCATIONS:
Overall Officials: Christian U. Blank, Prof., Principal Investigator — Medical oncologist/researcher
Locations (1):
- Antoni van Leeuwenhoek ziekenhuis, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Rozeman EA, Versluis JM, Sikorska K, Hoefsmit EP, Dimitriadis P, Rao D, Lacroix R, Grijpink-Ongering LG, Lopez-Yurda M, Heeres BC, van de Wiel BA, Flohil C, Sari A, Heijmink SWTPJ, van den Broek D, Broeks A, de Groot JWB, Vollebergh MA, Wilgenhof S, van Thienen JV, Haanen JBAG, Blank CU. IMPemBra: a phase 2 study comparing pembrolizumab with intermittent/short-term dual MAPK pathway inhibition plus pembrolizumab in patients with melanoma harboring the BRAFV600 mutation. J Immunother Cancer. 2023 Jul;11(7):e006821. doi: 10.1136/jitc-2023-006821. PMID 37479483